CLINICAL TRIAL: NCT02593344
Title: Peripheral Endothelial Function in Asthmatic Patients
Acronym: Endothasthm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/54
Record Dates: First submitted 2015-10-16; First posted 2015-11-02 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Endothelial Function
Keywords: asthma, endothelial function
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endopat (Experimental): measure of endothelial function with endopat
  Interventions: Device: Endopat

INTERVENTIONS:
Device: Endopat — measure of peripheral endothelial function by the reactive hyperemia-peripheral artery tone index with a specific device (Endopat)

SUMMARY:
The aim of the study is to assess the peripheral endothelial function in adult asthmatic patients and the relationship between the peripheral endothelial function and the pulmonary function.

DETAILED DESCRIPTION:
The primary criteria is the peripheral endothelial function that will be assessed by the measure of flow-mediated dilation (reactive hyperemia-peripheral artery tone index). The pulmonary function will be assessed by the measures of the FEV1, the forced vital capacity (FVC) and the expiratory flow between 25% and 75% (FEF25-75%). The relationship between these parameters of the pulmonary function and the peripheral endothelial function will be analyzed. In addition, a relationship between peripheral endothelial function and the level of asthma control (Asthma Control Test (ACT)), the cardiovascular risk factors (SCORE INdex) and the treatment for asthma (controllers) will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a clear-cut history of asthma at the time of enrolment into the trial (eventually confirmed in the past and documented by an increased hyperresponsiveness to methacholine; or a bronchodilator reversibility to a beta-2-adrenergic drug).

Exclusion Criteria:

* Patients with unstable asthma
* Patients with a significant acute disease other than asthma. A significant disease is defined as a disease which, in the opinion of the investigator, may influence the results of the trial.
* Pregnant or nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2015-04-09 (Actual); Study Completion 2015-04-09 (Actual)

PRIMARY OUTCOMES:
measure of reactive hyperemia-peripheral artery tone index | day 1
  measure of reactive hyperemia-peripheral artery tone index

SECONDARY OUTCOMES:
measure of the forced expiratory flow in one second (FEV1) | day 1
  measure of the forced expiratory flow in one second (FEV1)
measure of the forced vital capacity (FVC) | day 1
  measure of the forced vital capacity (FVC)
measure of expiratory flow between 25% and 75% (FEF25-75%) | day 1
  measure of expiratory flow between 25% and 75% (FEF25-75%)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, MD PhD, Principal Investigator — Foch hospital
Locations (2):
- France (2):
  - Hôpital Saint Antoine, Pulmonary function test laboratory, Paris
  - Hôpital Foch Department of pneumology, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Lockette W, Otsuka Y, Carretero O. The loss of endothelium-dependent vascular relaxation in hypertension. Hypertension. 1986 Jun;8(6 Pt 2):II61-6. doi: 10.1161/01.hyp.8.6_pt_2.ii61. PMID 3087875
- [Background] Ibengwe JK, Suzuki H. Changes in mechanical responses of vascular smooth muscles to acetylcholine, noradrenaline and high-potassium solution in hypercholesterolemic rabbits. Br J Pharmacol. 1986 Feb;87(2):395-402. doi: 10.1111/j.1476-5381.1986.tb10829.x. PMID 3955307
- [Background] Henno P, Boitiaux JF, Douvry B, Cazes A, Levy M, Devillier P, Delclaux C, Israel-Biet D. Tobacco-associated pulmonary vascular dysfunction in smokers: role of the ET-1 pathway. Am J Physiol Lung Cell Mol Physiol. 2011 Jun;300(6):L831-9. doi: 10.1152/ajplung.00251.2010. Epub 2011 Mar 4. PMID 21378026
- [Background] Peinado VI, Barbera JA, Ramirez J, Gomez FP, Roca J, Jover L, Gimferrer JM, Rodriguez-Roisin R. Endothelial dysfunction in pulmonary arteries of patients with mild COPD. Am J Physiol. 1998 Jun;274(6):L908-13. doi: 10.1152/ajplung.1998.274.6.L908. PMID 9609729
- [Background] Hughes R, Tong J, Oates C, Lordan J, Corris PA. Evidence for systemic endothelial dysfunction in patients and first-order relatives with pulmonary arterial hypertension. Chest. 2005 Dec;128(6 Suppl):617S. doi: 10.1378/chest.128.6_suppl.617S. No abstract available. PMID 16373872
- [Background] Wolff B, Lodziewski S, Bollmann T, Opitz CF, Ewert R. Impaired peripheral endothelial function in severe idiopathic pulmonary hypertension correlates with the pulmonary vascular response to inhaled iloprost. Am Heart J. 2007 Jun;153(6):1088.e1-7. doi: 10.1016/j.ahj.2007.03.005. PMID 17540215
- [Background] Peled N, Bendayan D, Shitrit D, Fox B, Yehoshua L, Kramer MR. Peripheral endothelial dysfunction in patients with pulmonary arterial hypertension. Respir Med. 2008 Dec;102(12):1791-6. doi: 10.1016/j.rmed.2008.06.014. Epub 2008 Aug 3. PMID 18678478
- [Background] Dorfmuller P, Perros F, Balabanian K, Humbert M. Inflammation in pulmonary arterial hypertension. Eur Respir J. 2003 Aug;22(2):358-63. doi: 10.1183/09031936.03.00038903. PMID 12952274
- [Background] Friedman R, Mears JG, Barst RJ. Continuous infusion of prostacyclin normalizes plasma markers of endothelial cell injury and platelet aggregation in primary pulmonary hypertension. Circulation. 1997 Nov 4;96(9):2782-4. doi: 10.1161/01.cir.96.9.2782. PMID 9386137
- [Background] Christman BW, McPherson CD, Newman JH, King GA, Bernard GR, Groves BM, Loyd JE. An imbalance between the excretion of thromboxane and prostacyclin metabolites in pulmonary hypertension. N Engl J Med. 1992 Jul 9;327(2):70-5. doi: 10.1056/NEJM199207093270202. PMID 1603138
- [Background] Xu W, Kaneko FT, Zheng S, Comhair SA, Janocha AJ, Goggans T, Thunnissen FB, Farver C, Hazen SL, Jennings C, Dweik RA, Arroliga AC, Erzurum SC. Increased arginase II and decreased NO synthesis in endothelial cells of patients with pulmonary arterial hypertension. FASEB J. 2004 Nov;18(14):1746-8. doi: 10.1096/fj.04-2317fje. Epub 2004 Sep 13. PMID 15364894
- [Background] Schanen JG, Iribarren C, Shahar E, Punjabi NM, Rich SS, Sorlie PD, Folsom AR. Asthma and incident cardiovascular disease: the Atherosclerosis Risk in Communities Study. Thorax. 2005 Aug;60(8):633-8. doi: 10.1136/thx.2004.026484. PMID 16061703
- [Background] Iribarren C, Tolstykh IV, Eisner MD. Are patients with asthma at increased risk of coronary heart disease? Int J Epidemiol. 2004 Aug;33(4):743-8. doi: 10.1093/ije/dyh081. Epub 2004 May 6. PMID 15131088
- [Background] Takemura M, Matsumoto H, Niimi A, Ueda T, Matsuoka H, Yamaguchi M, Jinnai M, Muro S, Hirai T, Ito Y, Nakamura T, Mio T, Chin K, Mishima M. High sensitivity C-reactive protein in asthma. Eur Respir J. 2006 May;27(5):908-12. doi: 10.1183/09031936.06.00114405. PMID 16707391
- [Background] Zureik M, Benetos A, Neukirch C, Courbon D, Bean K, Thomas F, Ducimetiere P. Reduced pulmonary function is associated with central arterial stiffness in men. Am J Respir Crit Care Med. 2001 Dec 15;164(12):2181-5. doi: 10.1164/ajrccm.164.12.2107137. PMID 11751184
- [Background] Zureik M, Kauffmann F, Touboul PJ, Courbon D, Ducimetiere P. Association between peak expiratory flow and the development of carotid atherosclerotic plaques. Arch Intern Med. 2001 Jul 9;161(13):1669-76. doi: 10.1001/archinte.161.13.1669. PMID 11434800
- [Background] Ayer JG, Belousova EG, Harmer JA, Toelle B, Celermajer DS, Marks GB. Lung function is associated with arterial stiffness in children. PLoS One. 2011;6(10):e26303. doi: 10.1371/journal.pone.0026303. Epub 2011 Oct 25. PMID 22046271
- [Background] Onufrak S, Abramson J, Vaccarino V. Adult-onset asthma is associated with increased carotid atherosclerosis among women in the Atherosclerosis Risk in Communities (ARIC) study. Atherosclerosis. 2007 Nov;195(1):129-37. doi: 10.1016/j.atherosclerosis.2006.09.004. Epub 2006 Oct 10. PMID 17045272
- [Background] Cakmak A, Zeyrek D, Cece H, Erel O. The relationship between carotid intima media thickness and oxidative stress in asthmatic children. Asian Pac J Allergy Immunol. 2010 Dec;28(4):256-61. PMID 21337909
- [Background] Yildiz P, Oflaz H, Cine N, Genchallac H, Erginel-Unaltuna N, Yildiz A, Yilmaz V. Endothelial dysfunction in patients with asthma: the role of polymorphisms of ACE and endothelial NOS genes. J Asthma. 2004 Apr;41(2):159-66. doi: 10.1081/jas-120026073. PMID 15115168
- [Background] Hazarika S, Van Scott MR, Lust RM, Wingard CJ. Pulmonary allergic reactions impair systemic vascular relaxation in ragweed sensitive mice. Vascul Pharmacol. 2010 Nov-Dec;53(5-6):258-63. doi: 10.1016/j.vph.2010.09.005. Epub 2010 Oct 1. PMID 20888432
- [Background] Heitzer T, Schlinzig T, Krohn K, Meinertz T, Munzel T. Endothelial dysfunction, oxidative stress, and risk of cardiovascular events in patients with coronary artery disease. Circulation. 2001 Nov 27;104(22):2673-8. doi: 10.1161/hc4601.099485. PMID 11723017
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Asmar R, Benetos A, Topouchian J, Laurent P, Pannier B, Brisac AM, Target R, Levy BI. Assessment of arterial distensibility by automatic pulse wave velocity measurement. Validation and clinical application studies. Hypertension. 1995 Sep;26(3):485-90. doi: 10.1161/01.hyp.26.3.485. PMID 7649586
- [Background] Hayward CS, Kraidly M, Webb CM, Collins P. Assessment of endothelial function using peripheral waveform analysis: a clinical application. J Am Coll Cardiol. 2002 Aug 7;40(3):521-8. doi: 10.1016/s0735-1097(02)01991-5. PMID 12142121
- [Background] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169
- [Background] Flammer AJ, Anderson T, Celermajer DS, Creager MA, Deanfield J, Ganz P, Hamburg NM, Luscher TF, Shechter M, Taddei S, Vita JA, Lerman A. The assessment of endothelial function: from research into clinical practice. Circulation. 2012 Aug 7;126(6):753-67. doi: 10.1161/CIRCULATIONAHA.112.093245. PMID 22869857
- [Background] Selamet Tierney ES, Newburger JW, Gauvreau K, Geva J, Coogan E, Colan SD, de Ferranti SD. Endothelial pulse amplitude testing: feasibility and reproducibility in adolescents. J Pediatr. 2009 Jun;154(6):901-5. doi: 10.1016/j.jpeds.2008.12.028. Epub 2009 Feb 12. PMID 19217124
- [Background] Dhindsa M, Sommerlad SM, DeVan AE, Barnes JN, Sugawara J, Ley O, Tanaka H. Interrelationships among noninvasive measures of postischemic macro- and microvascular reactivity. J Appl Physiol (1985). 2008 Aug;105(2):427-32. doi: 10.1152/japplphysiol.90431.2008. Epub 2008 May 15. PMID 18483158
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Mahmud FH, Van Uum S, Kanji N, Thiessen-Philbrook H, Clarson CL. Impaired endothelial function in adolescents with type 1 diabetes mellitus. J Pediatr. 2008 Apr;152(4):557-62. doi: 10.1016/j.jpeds.2007.08.044. Epub 2007 Nov 5. PMID 18346515
- [Background] Lowenstein L, Damti A, Pillar G, Shott S, Blumenfeld Z. Evaluation of endothelial function in women with polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2007 Oct;134(2):208-12. doi: 10.1016/j.ejogrb.2007.02.011. Epub 2007 Mar 19. PMID 17374431
- [Background] Roifman I, Sun YC, Fedwick JP, Panaccione R, Buret AG, Liu H, Rostom A, Anderson TJ, Beck PL. Evidence of endothelial dysfunction in patients with inflammatory bowel disease. Clin Gastroenterol Hepatol. 2009 Feb;7(2):175-82. doi: 10.1016/j.cgh.2008.10.021. Epub 2008 Oct 30. PMID 19121648
- [Background] Itzhaki S, Lavie L, Pillar G, Tal G, Lavie P. Endothelial dysfunction in obstructive sleep apnea measured by peripheral arterial tone response in the finger to reactive hyperemia. Sleep. 2005 May;28(5):594-600. doi: 10.1093/sleep/28.5.594. PMID 16171272